CLINICAL TRIAL: NCT03247101
Title: Probiotics for Gallstones in Post-bariatric Surgery Patients：A Prospective
Brief Title: Probiotics for Gallstones in Post-bariatric Surgery Patients：A Prospective Randomized Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Min-Sheng General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MSIRB2016006
Record Dates: First submitted 2017-08-08; First posted 2017-08-11 (Actual); Last update posted 2017-08-11 (Actual); Status verified 2016-08

CONDITIONS: Clostridium Butyricum Miyairi; Gallstones; Gastrointestinal Quality of Life Index
MeSH Terms: conditions — Gallstones

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Probiotics group (Experimental): Miyarisan-BM (Clostridium Butyricum Miyairi) 40 mg po tid x 6 months
  Interventions: Drug: Miyarisan-BM (Clostridium Butyricum Miyairi)
- Urso group (Active Comparator): ursodoxycholic acid, 200mg po tid x 6 months
  Interventions: Drug: Urso group
- Biotase group (Active Comparator): Biotase 1# [Biodiastase 30mg + lipase 65mg + newlase 10mg]/tab po tid x 6 months
  Interventions: Drug: Biotase group

INTERVENTIONS:
Drug: Miyarisan-BM (Clostridium Butyricum Miyairi) — 40mg po tid x 6months
  Arms: Probiotics group
Drug: Urso group — ursodoxycholic acid, 200mg po tid x 6 months
  Arms: Urso group
Drug: Biotase group — Biotase 1# [Biodiastase 30mg + lipase 65mg + newlase 10mg]/tab po tid x 6 months
  Arms: Biotase group

SUMMARY:
Morbid obesity has become a major global health problem, and the use of bariatric surgery is increasing. One common complication seen following bariatric surgery is the formation of gallstones. Contributing factors to gallstone formation include hypomotility of gall bladder and supersaturation of bile due to rapid weight loss and mobilization of cholesterol. Previous studies revealed oral probiotics could reduce the cholesterol level by as much as 22% to 33%. The possible mechanisms included bile salt hydrolase activity, assimilation of cholesterol by the bacteria, binding of cholesterol to the bacterial cell wall and physiological actions of the end products of short chain fatty acid fermentation. Therefore, the aim of this study was to determine the ability of probiotics to prevent gallstones formation after bariatric surgery and to evaluate the impact of oral administration of probiotics on the post bariatric surgery patients 's quality of life.

Gastrointestinal Quality of Life Index is a widely accepted questionnaire for evaluating the quality of life for patients receiving bariatric surgery. It consists of five domains: digestive symptoms; physical function; emotional condition; social condition and effect of medical treatment, which could access the quality of life of bariatric patient effectively and completely.

ELIGIBILITY:
Inclusion Criteria:

1. Patients receiving bariatric surgery for morbid obesity
2. Patiets at ages between 20 to 65 y/o
3. Patients willing to follow up regulary after bariatric surgery.

Exclusion Criteria:

1. Patients having gallstones before bariatric surgery
2. Patients refusing taking probiotics or refusing regular follow up after bariatric surgery

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2016-02; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Gallstones formation | 6 months

SECONDARY OUTCOMES:
serum total cholesterol and LDL level | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Min sheng general hospital, Taoyuan, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Shiffman ML, Sugerman HJ, Kellum JM, Brewer WH, Moore EW. Gallstone formation after rapid weight loss: a prospective study in patients undergoing gastric bypass surgery for treatment of morbid obesity. Am J Gastroenterol. 1991 Aug;86(8):1000-5. PMID 1858735
- [Result] Shiffman ML, Sugerman HJ, Kellum JH, Brewer WH, Moore EW. Gallstones in patients with morbid obesity. Relationship to body weight, weight loss and gallbladder bile cholesterol solubility. Int J Obes Relat Metab Disord. 1993 Mar;17(3):153-8. PMID 8385075
- [Result] Shiffman ML, Sugerman HJ, Kellum JM, Moore EW. Changes in gallbladder bile composition following gallstone formation and weight reduction. Gastroenterology. 1992 Jul;103(1):214-21. doi: 10.1016/0016-5085(92)91115-k. PMID 1612328
- [Result] Williams C, Gowan R, Perey BJ. A Double-Blind Placebo-controlled Trial of Ursodeoxycholic Acid in the Prevention of Gallstones during Weight Loss after Vertical Banded Gastroplasty. Obes Surg. 1993 Aug;3(3):257-259. doi: 10.1381/096089293765559278. PMID 10757929
- [Result] Worobetz LJ, Inglis FG, Shaffer EA. The effect of ursodeoxycholic acid therapy on gallstone formation in the morbidly obese during rapid weight loss. Am J Gastroenterol. 1993 Oct;88(10):1705-10. PMID 8213711
- [Derived] Han ML, Lee MH, Lee WJ, Chen SC, Almalki OM, Chen JC, Wu CC. Probiotics for gallstone prevention in patients with bariatric surgery: A prospective randomized trial. Asian J Surg. 2022 Dec;45(12):2664-2669. doi: 10.1016/j.asjsur.2022.01.120. Epub 2022 Feb 26. PMID 35232647